CLINICAL TRIAL: NCT04153851
Title: Effect of Neurectomy of Nasopalatine Nerve on Sensation of Anterior Palate in Patient Undergoing Rehabilitation of Atrophic Anterior Maxillary Ridge With Dental Implant
Brief Title: Study the Effect of Neurectomy of Nasopalatine Nerve on Sensation of Anterior Palate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed hamdi morsi, Principle investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: OMFS 6-3-1
Record Dates: First submitted 2019-11-02; First posted 2019-11-06 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Missing Teeth
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neurectomy of nasopalatine nerve (Other): 1. Prophylactic preoperative antibiotic will be administered prior to surgery.
  2. Oral disinfection will be performed before surgery.
  3. Labial infiltration anesthesia and nasopalatine nerve block anasthesia.
  4. The nasopalatine foramen will be exposed after reflection of a palatal and buccal flap.
  5. Severing of nerurovascular bundle and pushing the nasopalatine canal content nasally and insertion of bone graft in the canal.
  6. Dental implant will be inserted in the central incisor location.
  Interventions: Procedure: neurectomy of nasopalatine nerve

INTERVENTIONS:
Procedure: neurectomy of nasopalatine nerve — Severing of nerurovascular bundle and pushing the nasopalatine canal content nasally and insertion of bone graft in the canal. Dental implant will be inserted in the central incisor location

SUMMARY:
Study the effect of neurectomy of nasopalatine nerve on the sensation of anterior palate in patients undergoing rehabilitation of anterior maxillary ridge with dental implant

DETAILED DESCRIPTION:
Replacement of missing teeth in the anterior maxilla could be challenging if enlargement of the nasopalatine canal which is located in the midline of the palate posterior to the maxillary central incisors or ridge atrophy occur after tooth extraction. This could place the neurovascular content of the nasopaltine canal in the path of the dental implant which may lead to complications such as nasopalatine canal cyst, sensory dysfunction or implant failure. Technique to overcome this problem have evolved including neurectomy of the nasopalatine canal content and obliteration of canal with bone graft.

Loss of sensation in anterior palate following this procedure could be an annoying complication for patients. In recent studies regaining of sensation following such procedure have been reported, Confirmation of such results is essential to rule out the side effect of loss of sensation in the anterior palatal region

ELIGIBILITY:
Inclusion Criteria:

* • Adult patients requiring dental implants placement in the anterior region of maxilla and has insufficient horizontal bone .

  * Patients should be free from any systemic conditions that may affect soft tissue healing.

Exclusion Criteria:

* • Patients with systematic disease that may complicate healing.

  * Uncontrolled diabetic patient.
  * Patients with advanced osteoporosis.
  * Patients under bisphosphonates treatment.
  * Patients with neurological disorders (neuralgias, Parkinson's disease).
  * Patients with horizontal ridge atrophy (if the horizontal dimension of the residual ridge <3mm as determined with ridge callipers).
  * Heavy smoker patients.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
two point discrimination test | six months
  This test will be performed using a calliper, the two points of the calliper are opened progressively in 1mm increments and care should be taken that the two points are touching the mucosa in the same time until the patient can discriminate two points of contact at which the distance between the two points is recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt